CLINICAL TRIAL: NCT00681837
Title: Prevalence of Gastroesophageal Reflux During Childhood and Teenage Years in France
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Paula Fernstrom, AstraZeneca
Other Study IDs: NIS-GFR-DUM-2008/1
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Gastroesophageal Reflux
Keywords: gastroesophageal reflux; prevalence; childhood; France
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: children from 0 to 17 years old

SUMMARY:
The purpose of this study is to assess prevalence of gastrooesophageal reflux during childhood and teenage years in France and to describe patients'symptoms and gastrooesophageal reflux management

ELIGIBILITY:
Inclusion Criteria:

* children from 0 to 17years old seen in consultation

Exclusion Criteria:

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children recruited by both GPs and paediatricians
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2008-05; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
assess prevalence of gastrooesophageal reflux during childhood and teenage years in France, particularly 0-1 year-old prevalence and 1-11 year-old prevalence | At the end of the study

SECONDARY OUTCOMES:
describe patients'symptoms and gastrooesophageal reflux management | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GOTTRAND, Study Chair — CHRU Lille - France; Geneviève BONNELYE, Principal Investigator — TNS Healthcare 92120 Montrouge - France
Locations (25):
- China (25):
  - Research Site, Hefei, Anhui
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Xiamen, Guangdong
  - Research Site, Zhongshan, Guangdong
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Jinan, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Ningbo, Zhejiang
  - Research Site, Rui’an, Zhejiang
  - Research Site, Wenzhou, Zhejiang